CLINICAL TRIAL: NCT02420626
Title: Volcano Crux Vena Cava Filter Registry
Brief Title: Evaluation of the Short and Long Term Performance and Clinical Outcomes of the Crux Vena Cava Filter System
Status: Withdrawn | Type: Observational
Why Stopped: An industry-wide, alternative, post-market study has been initiated
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 140203
Record Dates: First submitted 2015-04-07; First posted 2015-04-20 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism; Deep Vein Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Crux Vena Cava Filter (VCF) Registry is a clinical study, sponsored by Volcano Corporation, to evaluate the short and long term performance and clinical outcomes of the Crux Vena Cava Filter System.

DETAILED DESCRIPTION:
The Crux VCF Registry is a non-randomized clinical study, sponsored by Volcano Corporation, to evaluate the short and long term performance and clinical outcomes of the Crux VCF System. The registry includes consecutive patients treated with the Crux VCF in a post-market (commercial) setting with data collection at the implant procedure through 2 years post implant or to filter retrieval, whichever comes first. Patients may also be enrolled (roll-in) from a previous Crux VCF implant within the previous 6 months. Follow up assessment will be performed at 6, 12 and 24 months post-implant and at the time of retrieval, if performed.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is >18 years of age.
2. Patient or their legally authorized representative understands the research nature of the study and is willing and capable of providing informed consent.
3. Scheduled for and receives a Crux VCF implant or;
4. Have previously had a Crux VCF implanted within the previous 6 months.

Exclusion Criteria:

1. Patient is scheduled for filter implant, but did not have a Crux VCF filter implanted due to anatomical exclusions or technical failures.
2. Patients unwilling or unable to comply with the protocol and provide informed consent.
3. Female patient of childbearing potential who is pregnant (she must have negative pregnancy test within the 48 hours prior to implantation and any retrieval procedure)
4. Patient is participating in another device or drug clinical trial that interferes with this protocol follow up schedule.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eligible for inclusion if they are scheduled for a vena cava filter implant with the Crux VCF System or have had a Crux VCF implanted within the previous 6 months for any of the following situations:
  1. Pulmonary thromboembolism when anticoagulation therapy is contraindicated;
  2. Failure of anticoagulation therapy in thromboembolic disease;
  3. Emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced; and
  4. Chronic, recurrent pulmonary embolism where anticoagulant therapy has failed or is contraindicated.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Prevention of Pulmonary Embolism | 2 years
  The primary objective is to evaluate the long term clinical outcomes of patients treated with the Crux VCF for the prevention of PE over a two year period or up to filter retrieval, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northside Vascular Surgery, Atlanta, Georgia
  - Rex Healthcare, Raleigh, North Carolina
  - Turkey Creek Medical Center, Knoxville, Tennessee